CLINICAL TRIAL: NCT00746395
Title: Randomized, Placebo-controlled Trial of Lubiprostone as a Preparation for Capsule Endoscopy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of South Alabama (Other)
Collaborators: Takeda (Industry); Sucampo Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 07-096
Record Dates: First submitted 2008-09-03; First posted 2008-09-04 (Estimated); Results first posted 2017-01-04 (Estimated); Last update posted 2020-10-08 (Actual); Status verified 2020-09

CONDITIONS: Inflammatory Bowel Disease
Keywords: capsule; endoscopy; prokinetic; lubiprostone; Normal; volunteers
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Lubiprostone; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- lubiprostone 24mcg single dose (Active Comparator): lubiprostone 24mcg single dose po prior to capsule endoscopy
  Interventions: Drug: Lubiprostone
- Sugar pill (Placebo Comparator): Placebo (sugar pill) - matched single dose po prior to capsule endoscopy
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lubiprostone — 24 mcg oral administration
  Other Names: Amitiza
  Arms: lubiprostone 24mcg single dose
Drug: Placebo — Oral administration
  Other Names: Sugar pill
  Arms: Sugar pill

SUMMARY:
This investigation is designed to compare lubiprostone and placebo for cleansing and propulsion in preparation for capsule endoscopy.

DETAILED DESCRIPTION:
Introduction of small bowel capsule endoscopy made available an unique technique for diagnostic evaluation of the gastrointestinal tract. After esophagogastroduodenoscopy and colonoscopy about 5% of bleeding cases remain unexplained and capsule endoscopy provides small bowel yield. Capsule endoscopy has special application for evaluation of inflammation bowel disease and other small bowel conditions. Several adjuncts are used to enhance the examination by improving cleansing preparation or propulsion. Metoclopramide, tegaserod, simethicone, erythromycin, phosphates and polyethylene glycol (PEG) colon cleansing agents have been tried and some show improved visualization or increased propulsion where more capsules reach to colonic cecum while still recording within the limits of its 8 hour battery. Recently, our group had an observational report of our experience showing that either full bowel cleansing preparation or prokinetics such as metoclopramide or tegaserod enhanced visualization and functioning capsule transit to the colon. Lubiprostone is a novel chloride channel activator that increases intestinal fluid secretion and motility. It is FDA approved and indicated for treatment of chronic idiopathic constipation.

This investigation is designed to compare lubiprostone and placebo for cleansing and propulsion in preparation for capsule endoscopy. The FDA approved 24 mcg constipation dose was chosen because other medications used in similar single dose in our pilot studies appear effective.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers

Exclusion Criteria:

* Gi disorders, gi surgery, cardiac, renal, or hepatic insufficiency, severe diarrhea

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2008-04; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: JAck A DiPalma, MD, Principal Investigator — University of South Alabama
Locations (1):
- USA Pavilion at Infirmary West, Mobile, Alabama, United States

REFERENCES:
- [Derived] Hooks SB 3rd, Rutland TJ, Di Palma JA. Lubiprostone neither decreases gastric and small-bowel transit time nor improves visualization of small bowel for capsule endoscopy: a double-blind, placebo-controlled study. Gastrointest Endosc. 2009 Nov;70(5):942-6. doi: 10.1016/j.gie.2009.04.045. Epub 2009 Jul 4. PMID 19577749

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruited from a specialty clinic in Mobile, AL, USA between April 2008 and September 2008.
Pre-assignment Details: 45 participants recruited and screened, 1 excluded, 4 withdrew from study.
Period: Overall Study
Arm/Group | Lubiprostone 24mcg Single Dose | Sugar Pill
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lubiprostone 24mcg Single Dose | Sugar Pill | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 40
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.75 (13.15045) | 35.4 (10.86472) | 37.07 (2.36881)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 12 | 27
  Male | 5 | 8 | 13
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Complete Small Bowel Transit
Description: Percent of subjects with capsule passage through small bowel
Time Frame: 8 hours
Population: Placebo 95%, lubiprostone 75%
Measure: Number; unit: percentage of subjects with passage
Arm/Group | Lubiprostone 24mcg Single Dose | Sugar Pill
Number analyzed (Participants) | 20 | 20
percentage of subjects with passage | 75 | 95

2. Secondary Outcome: Small Bowel Transit
Description: Small bowel transit time
Time Frame: Duration of the test - 8 hours
Population: Patients without transit to cecum were excluded
Measure: Mean (Standard Error); unit: Minutes
Arm/Group | Lubiprostone 24mcg Single Dose | Sugar Pill
Number analyzed (Participants) | 15 | 19
Minutes | 188.1 (68.0) | 218.9 (89.0)

ADVERSE EVENTS:
Time Frame: From the administration of the drug through the end of the procedure.
Description: No serious adverse events during study duration
Arm/Group | Lubiprostone 24mcg Single Dose | Sugar Pill
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 1/20 | 1/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lubiprostone 24mcg Single Dose (N=20) | Sugar Pill (N=20)
Headache (General disorders) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
Study participant enrollment met per protocol requirement.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes